CLINICAL TRIAL: NCT06100159
Title: Short-term Effects of Ventilation Tubes in Children With Chronic Otitis Media With Effusion Treated in ENT Private Practice; a Randomised Controlled Trial
Brief Title: Short-term Effects of Ventilation Tubes in Children With Chronic Otitis Media With Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Danish Medical Association (Other)
Responsible Party: Principal Investigator, Preben Homøe, Professor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REG-131-2015
Record Dates: First submitted 2017-02-17; First posted 2023-10-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Otitis Media With Effusion in Children; Quality of Life; Sleep
MeSH Terms: interventions — Middle Ear Ventilation

STUDY DESIGN:
Intervention Model Description: RCT with an intervention and a control group
Who Masked: Outcomes Assessor
Masking Description: questionnaires and sleep outcome measures will be assessed by masked person
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tympanostomy tube (Experimental): Insertion of tympanostomy tubes after 3 months observation for chronic otitis media with effusion (OME) according to the National guidelines in Denmark. Sleep measurements with accelerometer 7 nights before and 7 nights after intervention. Caregivers report use of paracetamol during nights with sleep measurements.
  Interventions: Device: Tympanostomy tube insertion
- Control (No Intervention): No tympanostomy tube treatment up to 1 month after enrollment in control group. Sleep measurements with accelerometer 7 nights at time of inclusion. Caregivers report use of paracetamol during nights with sleep measurements.
  After 1 month tympanic tube insertion is allowed if still chronic OME. If tympanostomy tubes are needed the children will undergo same evaluation as the intervention group.

INTERVENTIONS:
Device: Tympanostomy tube insertion — Ventilation tube insertion in the tympanic membrane
  Other Names: ventilation tube; grommet
  Arms: Tympanostomy tube

SUMMARY:
The goal of this clinical, randomized trial is to compare the sleeping patterns and quality of life of children with chronic otitis media with effusion (OME) with or without tympanic tubes insertion. The main questions it aims to answer are:

* Does tympanic tube insertion have an effect on sleep quality in children with chronic OME?
* Does tympanic tube insertion improve the quality of life for the children with chronic OME and their caregivers?

Participants will have their movements during sleep and number of awakenings measured by an accelerometer placed on their wrist for 7 nights before and after tympanic tube insertion. Their caregivers will answer questionnaires regarding quality of life on behalf of the child. Researchers will compare with a control group of children who also is diagnosed with chronic OME. They will also have their sleep monitored for 7 nights and their caregivers will complete quality of life questionnaires, but the will not receive a tympanic tube. However the control group will be reassessed a month after baseline, and if they still qualify for tympanic tube insertion they will undergo the same routine as the intervention group.

DETAILED DESCRIPTION:
Statement of intent

Background Otitis media with effusion (OME) is a common condition in the population of young children in Denmark. Sixty percent of the Danish children will experience at least one episode of OME or acute otitis media before they are 7 years old.

OME is a condition defined by non-purulent inflammation of the middle ear with serous and/or mucinous secretion why it is also known as serous otitis media. The diagnosis is most often made by a general practitioner or an ear nose-throat (ENT) specialist by otoscopy and measuring the middle ear pressure with a tympanometer. After a period of 3 months with persistent fluid in the middle ear, the treatment is usually insertion of a tympanostomy tube, also called a grommet, in the tympanic membrane. OME may be accompanied by varying degrees of non-infectious symptoms, including earaches, hearing loss and reduced quality of life.

Tympanostomy tube insertions (TTI) are also performed in children with recurring acute otitis media. The Danish Health Authority, "Sundhedsstyrelsen", has collaborated with multiple Danish ENT specialists and published a peer reviewed National Clinical Guideline (NCG) regarding TTI.

Denmark has the highest rate of tympanostomy tube insertion (TTI) in children in the world. Every year around 36.000 TTI are performed on children in Denmark. The annual incidence is 108 : 1.000 for children between 0-3 years of age and 35 : 1.000 in children between 0-15 years of age. In comparison, the annual incidence is lower than 10 : 1.000 in United Kingdom, USA and Canada. Recent studies by DØNHOF (Danish Ear-, Nose, and Throat Specialists Organization Research Group) have shown that the vast majority of TTI procedures are conducted according to the National Clinical Guidelines (NCG).

However, this major difference in procedure ratio between countries raises questions. Is the procedure performed too often in Denmark or not often enough in other countries? Do more children suffer from OME in Denmark compared to other parts of the world? Large and thorough studies have been made to assess the impact of TTI on hearing, speech and cognitive development of children with OME. So far has no significant, long-term benefits been found.

High quality studies on quality of life (QoL) in children with OME and their caregivers are few. Questionnaire studies on this subject find that caregivers generally report improved QoL for their children after TTI. In particular, the caregivers describe a poor and broken-up sleep pattern when their child is diagnosed with OME. They also report that the sleep pattern significantly improves after TTI, which increases QoL for the child as well as their caregivers. These QoL questionnaire studies have not been randomized and are at high risk of selection bias where caregivers may prefer TTI.

Even the most recent, nationally published studies have pointed out the need for an objective, randomized evaluation of the effect of TTI. This has not been possible until recently.

New FDA-approved technology, the Actigraph gt3x+ 3-axis accelerometer makes it possible to objectively register movement during sleep, awakenings and total amount of sleep and thereby evaluate the quality of the children's sleep, also called sleep efficiency.

It is internationally discussed how long an observation period for OME is needed before treatment with TTI is indicated. In Denmark and many other countries, the period of observation is set to 3 months. An observational patient reported outcome (PRO) study by caregivers to children offered TTI from 26 ENT clinics spread across Denmark showed that 91% of TTI procedures were conducted adherent to the NCG. However, this was without data on hearing loss or tympanometry. OME is a condition that can be resolved spontaneously, so if you apply a longer observation period, it is possible, that fewer children would undergo surgery. Therefore there is a need to study if the current NCG is of benefit for the children and their families compared to a longer observation period.

Objectives

1. Evaluate the sleep efficiency of children with OME before and after TTI by state-of the-art objective measurement using the Actigraph gt3x+ accelerometer and a validated questionnaire. The decision to perform TTI will be in accordance with the NCG.
2. Evaluate the children's and their caregiver's QoL before and after TTI through validated questionnaires and measurements of the children's sleep pattern.
3. Evaluate if the currently recommended observation period of 3 months is sufficient, or if 4 months observation would be more appropriate.

Hypotheses

1. TTI in children with OME induces better sleep patterns and better sleep efficiency.
2. The children and their caregiver's QoL is improved by TTI.
3. The current observation period of 3 months before deciding on TTI is satisfactory.

Methods Study design The study design is a randomized controlled trial. The person analyzing the sleep efficiency will be blinded to the randomization, not knowing if the data is coming from the intervention or the control group. For ethical and practical reasons the caregivers and children cannot be blinded to the randomization.

The majority of TTI surgery in Denmark is performed by private practicing ear-nose-throat (ENT) specialists as a part of the public health facilities. The ENT specialist will be responsible for including the children when they meet the requirements of the NCG for the TTI procedure and screen for the exclusion criteria. The children must be diagnosed with OME for three consecutive months, and the caregivers suspect that their child's hearing is impaired. If the child matches the inclusion criteria, they and their caregivers will be informed about the trial verbally and in writing before they are asked to join. The children are included longitudinally and will be randomized into the intervention or the control group.

The intervention group will be scheduled for TTI performed by the ENT specialist as per NCG with sleep registration 7 nights before and after the procedure. The control group will go through a 7-night sleep registration at the inclusion point and then an additional month of observation. Afterwards the children in the control group will be reassessed by the ENT specialist. If they still meet the inclusion criteria for TTI, they will be offered the procedure and will be included in the intervention group. For both groups, the ENT specialist must fill out the provided questionnaires, documenting the caregiver reported symptoms before TTI and the objective findings including otomicroscopy and tympanometry before and after the TTI. The impact of TTI on hearing has been thoroughly investigated and is therefore not an end outcome in this study. However, questions regarding the caregiver's assessment of changes in the child's hearing is included in the questionnaires. The QoL questionnaires for the caregivers are to be answered at time of inclusion and, depending on the group, again after TTI or again after 1 month of observation.

The caregivers are asked to write down the time their child was put to bed, if they provided their child with paracetamol at any time and estimate how long their child slept each night. There will also be an option to comment on if there were any competing illnesses in the period of sleep registration.

To register the children's activity in their sleep, and thereby their sleeping pattern and efficiency, they will be fitted with a 3-axis accelerometer called the Actigraph gt3x+, which in shape and size resembles a wristwatch. It is a noninvasive monitor, which provides precise and validated data about movement during sleep. It is an FDA approved medico-technical equipment and state-of-the-art for measuring activity in children. The children will wear the watch on their wrist at nighttime only.

The children's sleep will be registered as close to the time of inclusion as possible, and exactly the 7 nights before the TTI and the 7 nights immediately after the procedure, which means 14 nights in total for the intervention group.

In the control group, their sleep will be monitored 7 nights at the time of the inclusion. After 1 month of observation they will be reassessed by the ENT specialist. If they still meet the criteria of the NCG they too will be offered TTI. If they accept, they will join the intervention group with the measurements of activity during sleep 7 nights before and 7 nights after TTI and the caregivers will again fill out the questionnaires. This sum up to a maximum of 21 nights with measurement in total for the children in the control group. Grommets of the type Donaldson will be used in all TTI procedures.

Research biobank In relation to this project there will be established a biobank. During a TTI procedure, the fluid in the middle ear is removed by suction to minimize risk of inflammation around and blockage of the ear tube/grommet. This fluid is normally discarded, but during this project, the fluid will be kept with the intention of later analysis for microbiome.

The analysis will include examination for bacteria and virus remnants, 16 s rRNA and 16 s rDNA. The fluid, which is comprised of about 2 mL per ear, is saved in an -80 degree Celsius freezer in the safe facilities.

The purpose of the biobank is to store the fluid until all samples are collected and the analysis tools are fully financed.

The biobank will cease to exist 31.12.2025. All excess fluids will be destroyed hereafter.

Statistical considerations The following mathematical assumptions were made to calculate the sample size. Estimated awakenings/periods of high activity during sleep before TTI: 6 episodes per night. Estimated reduced awakenings/periods of high activity during sleep = 20% meaning 6 x 0,8 = 4,8 episodes per night after TTI. The estimated standard deviation for the normal child population: 2-8 episodes per night.

The calculated standard deviation equals 8-2 = 6 x 0,95 = 5,70/4 = 1,425. Type 1 error (α) is set per standard 0,05. Type 2 error (β) is set per standard 0,2 and power is set to 0,8. The calculated sample size for each group equals 24 children, meaning 48 children in total.

Finally, a dropout rate of 20% is estimated and add that to our total: 48 x 1,2 = 58 children. Investigators has chosen to round that up to 60.

The sample size is as follows: 30 children in the control group and 30 children in the intervention group. Keeping in mind, that the 30 children in the control group can, after the 1 month of observation, also be included in the intervention group, if they still meet the NCG criteria for TTI. That means the potential of 60 children in the intervention group.

Scientific and socioeconomic perspectives Even the most up-to date national and international studies and reviews request randomized controlled studies investigating the effects of TTI. This randomized controlled study will provide completely new knowledge no matter the outcome. It is the first to measure sleep efficiency in relation to OME. If it proves a significant and objectively measured improvement in sleep after TTI, and it correlates to the answers in the QoL questionnaires, it could be an international game changer with benefits for the children suffering from OME and a support to the clinical practice in Denmark. A good sleep is such an important factor in a child's ability to acquire new knowledge and for their caregivers to be able to go to work and function at work. Therefore, it could lead to new international clinical guidelines for TTI and bring better QoL to the children with OME and their families. If our study does not show a significant effect that could give evidence to suggest a reduction in TTI among children in Denmark.

Side effects and risks to participants Partaking in this study will not cause any health risks to the participants compared to children that do not partake in the study. There are no documented side effects, complications, or disadvantages to waiting an additional month before getting TTI. (10) The overall risk associated with TTI are mainly the risks of general anesthesia and a 1-6% risk of a persisting perforation of the tympanic membrane, that could require surgical treatment. There are no risks involved in the usage or wearing of the Actigraph gt3x+ accelerometer, which is FDA approved. The Actigraph gt3x+ accelerometer has previously been used in numerous studies measuring activity of children.

Scientific ethical considerations This trial has been approved by the Danish Committee for Scientific Research ("Nationale Videnskabsetiske Komité") REG-131-2015 and meet the criteria of category C in their guideline's section 4.2.1.1. The trial has also been approved by The Danish Data Protection Agency "Datatilsynet" and is registered on clinicaltrials.gov. Information about the participants is protected by The General Data Protection Regulation (GDPR).

Practical Feasibility This study was initiated by Principal investigator Preben Homøe, MD, Ph.d, DMSc and professor at the Department of Otorhinolaryngology and Maxillofacial Surgery, Zealand University Hospital, together with field researcher and colleague Trine Nybo Ranneries, MD. Two ENT specialists with each their own private ENT clinic (Peter Kofoed Tingsgaard, MD, PhD and Christian Hamilton Heidemann MD, PhD) have participated from the beginning of the planning of the study and acted as study sites with inclusion of patients, gathering of consent, questionnaires and performing the TTI and controls.

Trine N. Ranneries is currently a specialist registrar, with 1 year remaining in training to become an ENT specialist and has been amanuensis in Peter Tingsgaard's practice.

The inclusion of participants and collection of data was started with funding from "Foreningen af Danske Speciallægers forskningsfond" (The Research Fond for the Danish Private Practitioners) to acquire the wActisleep watches and software.

At present time, all 60 participants have been included and the follow-up period has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-4 years with chronic otitis media with effusion and subjective hearing loss
* 1. time ventilation tube insertion
* At least three months with middle ear fluid in both ears before inclusion
* ASA group 1 and 2

Exclusion Criteria:

* Recurrent AOM
* Concomitant adenoidectomy or adenotonsillectomy
* Lip-gum-cleft anomalies or other craniofacial malformations
* Downs syndrome
* Existing sleep apnea
* Asthmatic bronchitis or other chronic lung diseases like CF or other sleep disorders
* ASA > 2
* Children with hyperkinetic syndrome
* Present breastfeeding during night
* Not fluent in Danish language
* Other systemic diseases

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality | For the intervention group: 7 nights before and 7 nights after intervention. For the control group: 7 nights at time of inclusion.
  Sleep length and quality. An accelerometer is fitted on the participants and measures movement in 3 axis. The movement counts from the acclerometer will be processed by Sadeh's algorithm giving assessed minutes of total sleep, awakenings and sleep quality. The outcome will be assessed by a blinded investigator.
Change in Quality of Life | At inclusion and up to 2 months follow up
  Quality of life quantified by the validated questionnaire OM-6. 7-point Likert scale where 1 is no problem and 7 is extreme problem. The global NRS scales were 10 point scales with o = worst possible QoL and 10 = best possible QoL

SECONDARY OUTCOMES:
Use of pain reliever | For the intervention group: 7 nights before and 7 nights after intervention. For the control group: 7 nights at time of inclusion.
  use of weak pain reliever, paracetamol, self-reported by caregivers. Not an intervention. Participants in the intervention and control group decides their own use of pain reliever. We ask them to report if they have used paracetamol during the nights with acc3lererometer measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Preben Homoee, MD, Principal Investigator — Zealand University Hospital
Locations (2):
- Denmark (2):
  - Ørelægerne Fredericia, Fredericia
  - Peter Tingsgaard, Slagelse

IPD SHARING:
Plan to Share IPD: Yes
All results in database will be published anonymously after study termination